CLINICAL TRIAL: NCT02968017
Title: Variability in Middle Cerebral Artery Doppler Measurements in Uncomplicated Term Pregnancies.
Brief Title: Middle Cerebral Artery Doppler in Uncomplicated Term Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Boaz.Weisz, Professor of Fetal Medicine, Sheba Medical Center
Other Study IDs: 3571-16-SMC
Record Dates: First submitted 2016-11-13; First posted 2016-11-18 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Post Date
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MCA-PI: Measurement Middle cerebral artery pulsatility index

SUMMARY:
Doppler measurements in the Middle Cerebral Artery (MCA) is a part of the assessment for assessing fetal well-being in complicated pregnancy, including Intra Uterine Growth Retardation and Fetal Anemia.

The use of this Doppler measurement in uncomplicated term pregnancies is not a common practice due to lack of information. However, several studies use the MCA Pulsatility Index (PI) as part of the Cerebro-Placental-Ratio (CPR) measurment at term.

The purpose of this trial is to assess MCA Doppler variability in term, uncomplicated pregnancy.

DETAILED DESCRIPTION:
Measuring the resistance in the fetal middle cerebral artery (MCA) is an important factor in assessing fetal well-being. On its own, the Pulsatility Index (PI) in the MCA may indicate a decrease in fetal oxygenation. Furthermore, the PI measured in the Fetal MCA is an index parameter in the calculation of the Cerebro-Placental Ratio (CPR) used to evaluate whether there is an existing disturbance in the Placental-Umbilical and Feto-cerebral circulations. The CPR is a measurement that enables practitioners to predict the fetuses reaction to intrauterine hypoxemia. The CPR measurement is commonly used to evaluate small for gestational age (SGA) fetuses and to distinguish between constitutionally small fetuses and ones that suffer from placental insufficiency. For those who suffer from placental insufficiency, the CPR measurement is an aid in deciding the optimal time and mode of delivery.

Recently, researchers pondered if the CPR measurement may aid in predicting disturbance in fetal oxygenation during delivery. A number of studies have showed that appropriate for gestational age fetuses with abnormal CPR measurements may be susceptible to delivery complications in the same manner as fetuses who suffer from placental insufficiency. The question that is yet to be answered is whether the MCA measurement reliable in term pregnancies. This question arises due to the impression that the MCA measurement at term is highly variable, even when taken under optimal conditions.

The aim of this study is to evaluate the intra-observer variability in the MCA measurement under optimal conditions, in Uncomplicated Term Pregnancies.

ELIGIBILITY:
Inclusion Criteria:

Uncomplicated Term Pregnancies

Exclusion Criteria:

High Risk Pregnancies including placental insufficiency, intrauterine growth retardation or any maternal vascular disease.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Uncomplicated singleton pregnancies at 37-42 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Pulsatility index (Doppler measurements) in the middle cerebral artery | Full Term Pregnancies (37 to 42 weeks)
  Measurement MCA-PI Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Weisz, Prof, Principal Investigator — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: Undecided